CLINICAL TRIAL: NCT06942117
Title: Investigating the Effect of Caffeine Consumption on Speech Understanding in Noise in Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Merve MERAL ÇETİNKAYA, Assistant professor, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 41/2025; 1919B012442147 (Other Grant/Funding Number: The Scientific and Technological Research Council of Türkiye (TÜBİTAK))
Record Dates: First submitted 2025-04-14; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Approximately 280 grams of caffeine containing coffee is given.
  Interventions: Other: Experimental
- Placebo (Placebo Comparator): Decaffeinated coffee will be provided.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Experimental — Approximately 280 grams of caffeine containing coffee will be given
  Arms: Experimental
Other: Placebo — Decaffeinated coffee will be given.
  Arms: Placebo

SUMMARY:
Caffeine is a widely consumed substance worldwide and is often used to increase alertness and improve cognitive functions. Caffeine stimulates brain activity by binding to adenosine receptors, which increases alertness instead of sleepiness. Studies on the effects of caffeine on cognitive functions have shown that it improves basic cognitive functions such as attention, reaction time, and alertness, while a less pronounced effect is seen on sensory functions such as vision and hearing. However, no study has been found investigating the effect of caffeine consumption on understanding speech in noise. Understanding speech in noise is a skill that includes not only auditory functions but also cognitive functions. This skill is affected by cognitive elements such as selective attention and executive functions. In this context, it is thought that this study, which aims to examine the relationship between caffeine and understanding speech in noise, will contribute to the literature. 60 participants between the ages of 18-30 will be included in this study. Participants will consist of individuals without hearing loss (SSO<25 dB nHL), no history of neurological or psychological disorders, non-smokers, and those who do not use ototoxic drugs. Participants will be randomly divided into a placebo group that consumes decaffeinated coffee and a study group that consumes coffee containing 300 mg caffeine. The Turkish Matrix Test will be administered 30 minutes after coffee consumption. In addition, participants will be asked to keep a caffeine diary for one week to determine their daily caffeine consumption and will be asked to fill out the Caffeine Use Disorder Scale. Thus, they will be divided into low and high caffeine consumption groups and their speech understanding skills in noise will be compared.

ELIGIBILITY:
Inclusion Criteria:

* For both groups, it was planned to include individuals who had no hearing loss (SSO<25 dB nHL), no history of neurological or psychological disorders, were non-smokers, and did not use ototoxic drugs.

Exclusion Criteria:

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2025-09-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Turkish Matrix Test | Before and 30 minutes after drinking coffee
  The test will be administered using the Oldenburg Measurement Application (OMA) software. Using the adaptive procedure, the signal-to-noise ratio (SNR-50) at which the individual repeats the words correctly at 50% will be found. Accordingly, the noise will be given continuously, kept constant at 65 dB SPL throughout the test. The test will start at 0 dB signal-to-noise ratio (SNR). There are sentences consisting of 5 words in the test. If the participant repeats at least three of the five words presented to him/her correctly, the SNR will decrease and if he/she does not repeat at least three words correctly, the SNR will increase. A total of 20 sentences will be presented to the participants.

SECONDARY OUTCOMES:
Caffeine Use Disorder Scale | Before consuming caffeine.
  This scale, developed by Ágoston et al. (2018), consists of 10 items based on the nine criteria recommended for caffeine use disorder specified in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). The scale measures the severity of caffeine use symptoms in the last twelve months. As the scale score increases, caffeine use disorder symptoms also increase. Kaya et al. (2021) conducted the Turkish validity and reliability study of the scale. The total score that can be obtained from this scale varies between 10 and 40 and there is no reverse item. The questions are graded as "1=never, 2=sometimes, 3=often, 4=very often" and are interpreted as caffeine use disorder increases as the scale score increases. In the reliability analysis, Cronbach alpha internal consistency coefficient was found to be 0.86, and the intraclass correlation coefficient was found to be 0.83.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Aydin University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No